CLINICAL TRIAL: NCT00004396
Title: Studies in Porphyria III: Heme and Tin Mesoporphyrin in Acute Porphyrias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Purpose: Treatment
Other Study IDs: 199/13185; UTMB-96-476; UTMB-96-318; UTMB-FDR000710; UTMB-FDR001459
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Rare Diseases | interventions — heme arginate; tin mesoporphyrin

INTERVENTIONS:
Drug: heme arginate
Drug: tin mesoporphyrin

SUMMARY:
OBJECTIVES: I. Compare the efficacy of heme arginate, singly or in combination with tin mesoporphyrin, in lowering porphyrin precursors in patients with asymptomatic acute intermittent porphyria.

II. Evaluate and compare the safety and tolerability of these treatment regimens in this patient population.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is an unblinded, dose ranging study. Patients receive heme arginate alone or in combination with tin mesoporphyrin.

Patients receive tin mesoporphyrin IV as a single dose. Heme arginate is administered as a single intravenous infusion.

Patients are entered in cohorts of 4. Subsequent cohorts of 4 patients each receive escalating doses of tin mesoporphyrin in combination with 1 of 2 different dosages of heme arginate. Subjects must maintain a constant diet.

Patients experiencing adverse reactions are followed as clinically indicated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Documented acute intermittent porphyria in remission for at least 1 month
* Increased excretion of porphyrin precursors
* Absence of neurovisceral symptoms due to porphyria for at least 1 month

--Prior/Concurrent Therapy--

* At least 1 month since prior heme preparation therapy
* Concurrent medication for coexisting condition is allowed, as long as dose and pattern of administration is held constant during study

--Patient Characteristics--

* Renal: Urinary porphobilinogen excretion of at least 20 mg every 24 hours
* Other: Not pregnant Fertile female patients must use effective contraception during and at least 6 months before study At least 1 month since any symptoms of disease No concurrent acute hemorrhagic disorder such as: Gastrointestinal bleeding Intracerebral hemorrhage No known hypersensitivity to heme arginate, tin mesoporphyrin, another heme preparation, or related heme analogue No other condition that may increase risk to patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 1997-09

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - University of Texas Medical Branch, Galveston, Texas